CLINICAL TRIAL: NCT06552052
Title: A Retrospective and Prospective Natural History of Genetic Vasculopathies
Status: Recruiting | Type: Observational
Sponsor: Massachusetts General Hospital (Other)
Responsible Party: Principal Investigator, Patricia Musolino, MD PhD, Dr. Patricia L. Musolino, MD PhD, Principle Investigator, Massachusetts General Hospital
Other Study IDs: 2023P000821
Record Dates: First submitted 2024-01-04; First posted 2024-08-13 (Actual); Last update posted 2025-05-08 (Actual); Status verified 2025-05

CONDITIONS: Multisystemic Smooth Muscle Dysfunction Syndrome; ACTA2

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (4):
- Cohort 1 (29 days - 6 years of age): 1. Patient is between the ages of 29 days - 6 years old
  2. Confirmed ACTA2 pathogenic variant
  3. Available medical records since birth that permit documentation of disease characteristics and developmental milestone
  4. Have two parents and/or legal guardians who are English speaking and are able to read, understand, and sign the informed consent
  5. Able to tolerate travel to study site
- Cohort 2 (7 - 18 years of age): 1. Patient is between the ages of 7 - 18 years old
  2. Confirmed ACTA2 pathogenic variant
  3. Available medical records since birth that permit documentation of disease characteristics and developmental milestone
  4. Have two parents and/or legal guardians who are English speaking and are able to read, understand, and sign the informed consent
  5. Able to tolerate travel to study site
- Cohort 3 (19 - 99 years of age): 1. Patient is between the ages of 19 - 100 years old
  2. Confirmed ACTA2 pathogenic variant
  3. Available medical records since birth that permit documentation of disease characteristics and developmental milestone
  4. Patient, parent and/or legal guardian is English speaking is able to read, understand, and sign the informed consent
  5. Able to tolerate travel to study site
- Cohort 4 (Retrospective - All Ages): 1. Patient of any age, alive or deceased
  2. Confirmed ACTA2 pathogenic variant
  3. Available medical records since birth that permit documentation of disease characteristics and developmental milestone
  4. Patient, parent and/or legal guardian is English speaking and able to read, understand, and sign the informed consent

SUMMARY:
This study will combine retrospective review of medical records from patients with ACTA2 and ongoing collection of clinical data using standardized instruments and intervals on an observational basis from patients with ACTA2.

Patients in cohorts 1-3 will be asked to attend clinic visits in person per the schedule of events. At minimum, the medical records of patients with ACTA2 will be reviewed to record data on aspects of the disease, including disease characteristics and developmental milestones. The study is planned to enroll a total of 100 patients: 7 in cohort 1, 7 in cohort 2, and the remaining in cohorts 3 and 4.

This study is planned to study patients for at least 3 years with the option to continue as long as possible for assessment of disease progression. During their continued study participation, as patients age, they may move into the next cohort. Beyond 3 years the duration of the study with be determined by availability of funding from sponsors.

ELIGIBILITY:
Inclusion Criteria:

* Confirmed ACTA2 pathogenic variant
* Available medical records since birth that permit documentation of disease characteristics and developmental milestone
* Have two parents and/or legal guardians who are English speaking and are able to read, understand, and sign the informed consent
* Able to tolerate travel to study site

Exclusion Criteria:

* Patient does not meet the inclusion criteria
* Patient is currently pregnant

Min Age: 29 Days | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Children who have been diagnosed with a genetic vasculopathy, ACTA2 R179 for example.
Sampling Method: Probability Sample
Enrollment: 50 (Estimated)
Dates: Start 2024-05-08 (Actual); Primary Completion 2027-12 (Estimated); Study Completion 2028-07 (Estimated)

PRIMARY OUTCOMES:
Retrospectively define sequence and timing of vascular and non-vascular symptoms and disease progression | 3 Years
  1.1 Develop patient surveys and identify retrospective/existing clinical data sources for aggregation, harmonization, and analyses of outcomes and biomarkers to be compared to existing published data. 1.2. Identify modifiers of symptom progression in patients with MSMDS. 1.3 Correlate the degree of disease progression by systems in 40 patients (cross-sectional study) and construct an MSMDS Rating Scale to evaluate disease severity and progression in children. 1.4 Create case report forms based on previously known and developed surveys in 1.1. to allow for standardized prospective data collection (Outcome 2).
Prospectively assess the rate of change of vascular and non-vascular disease in MSMDS using quantitative measures, patient/caregivers reported outcomes (PROs). | 3 Years
  2.1 Assess vascular and non-vascular disease progression over 3 years. 2.2 Compare the trajectory between clinical rating scales and patient-reported outcomes. 2.3 Correlate disease progression by individual and MSMDS-specific scale with other variables (age at diagnosis, sex, genetic variance, surgeries, etc).
Determine whether remote assessments with wearable technology systems are comparable with quantitative performance measures obtained in Aim 2 | 3 Years
  Use the Actigraphy wearable technology system in conjunction with a video consult to remotely assess gait, limb movement and exercise performance.

CONTACTS AND LOCATIONS:
Locations (1):
- Massachusetts General Hospital, Boston, Massachusetts, United States

IPD SHARING:
Plan to Share IPD: No